CLINICAL TRIAL: NCT00145145
Title: Phase I/II Study of Immunization With the MAGE-3.A1 Peptide Mixed With the Immunological Adjuvant CpG 7909 in Patients With Metastatic Melanoma
Brief Title: Immunization With the MAGE-3.A1 Peptide Mixed With the Adjuvant CpG 7909 in Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2002-001
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; Vaccine; Peptide; MAGE; CpG
MeSH Terms: conditions — Melanoma | interventions — ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAGE-3.A1 Peptide mixed with CpG 7909 (Experimental): Patients were vaccinated every two weeks on six occasions. On each vaccination day, the MAGE-3.A1 peptide (300 mcg) mixed with CpG 7909 (5 mg) was administered twice intradermally (10% of the dose each) and twice subcutaneously (40% of the dose each) in the arms and thighs.
  Interventions: Biological: MAGE-3.A1 peptide and CpG 7909

INTERVENTIONS:
Biological: MAGE-3.A1 peptide and CpG 7909

SUMMARY:
The purposes of this study are to determine whether immunization with the MAGE-3.A1 peptide mixed with CpG 7909 results in a detectable immune response; to determine the safety of this vaccine and to document the tumor response to the vaccine.

DETAILED DESCRIPTION:
Patients will be vaccinated every two weeks on six occasions. On each vaccination day, the MAGE-3.A1 peptide (300 µg) mixed with CpG 7909 (5 mg) will be administered twice intradermally (10% of the dose each) and twice subcutaneously (40% of the dose each) in the arms and thighs.

Tumor staging will be performed before inclusion and at week 13. PBL collections will be performed before starting the treatment, and at weeks 3, 7 and 13. They will provide the T lymphocytes for the immunological analysis.

Additional cycles of immunization will be proposed to patients without tumor progression requiring another treatment. A second cycle of 3 injections at 6-week intervals will be started at week 17 with the same vaccine, followed by a third cycle of 12 injections at 3-month intervals starting at month 11. At any time, progression of the disease necessitating any treatment not allowed during the study, will result in study withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven cutaneous melanoma, or clear cell sarcoma, which is considered as a subtype of melanoma.
2. Melanoma must be at one of the following AJCC 2002 stages:

   * Regional metastatic disease (any T; N2b, N2c or N3; M0).
   * Distant metastatic disease (any T; any N; M1a, M1b or M1c), except brain or leptomeningeal localizations, and except elevated LDH.
3. Patients must be HLA-A1.
4. Melanoma must express the MAGE-3 gene, as determined by RT-PCR.
5. Presence of at least one measurable or non-measurable tumor lesion, excluding leptomeningeal metastasis.
6. Expected survival of at least 3 months.
7. Karnofsky performance scale ≥70 or WHO performance status of 0 or 1.
8. Within the last 4 weeks prior to study day 1, vital laboratory parameters should be within normal range, except for the following laboratory parameters, which must be within the ranges specified:

   Lab Parameter Range
   * Hemoglobin ≥ 10 g/dl or ≥ 6,25 mmol/l
   * Granulocytes ≥ 1,500/µl
   * Lymphocytes ≥ 700/µl
   * Platelets ≥ 100,000/µl
   * Serum creatinine ≤ 2.0 mg/dl or ≤ 177 µmol/l
   * Serum bilirubin ≤ 2.0 mg/dl or ≤ 34.2 µmol/l
   * ASAT and ALAT ≤ 2 x the normal upper limits
   * LDH ≤ the normal upper limit.
9. Viral tests:

   * HIV (human immunodeficiency virus): negative antibodies.
   * HBV (hepatitis B virus): negative antigens; antibodies may be positive.
   * HCV (hepatitis C virus): negative antibodies.
10. Age ≥ 18 years.
11. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Previous treatment with more than one regimen of systemic chemotherapy, combined or not with non-specific immunotherapy such as interferon alpha or interleukins. Chemoimmunotherapy or radiotherapy must be stopped within the preceding 4 weeks (6 weeks for nitrosoureas and mitomycin C).
2. Previous treatment with a vaccine known or likely to contain the MAGE-3.A1 antigen, unless there is evidence that no CTL response against this antigen was induced by the vaccine.
3. Clinically significant heart disease i.e. NYHA class 3 congestive heart failure; myocardial infarction within the past six months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
4. Active immunodeficiency or autoimmune disease. Vitiligo is not an exclusion criterion.
5. Other serious acute or chronic illnesses, e.g. active infections requiring antibiotics, bleeding disorders, or other conditions requiring concurrent medications not allowed during this study.
6. Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
7. Lack of availability for immunological and clinical follow-up assessments.
8. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
9. Pregnancy or breastfeeding.
10. Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-01-12 (Actual); Primary Completion 2005-04-07 (Actual); Study Completion 2008-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas van Baren, MD, Study Chair — Ludwig Institute for Cancer Research; Thierry Boon, PhD, Study Director — Ludwig Institute for Cancer Research
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc (UCL), Brussels
  - Ludwig Institute for Cancer Research, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchand M, van Baren N, Weynants P, Brichard V, Dreno B, Tessier MH, Rankin E, Parmiani G, Arienti F, Humblet Y, Bourlond A, Vanwijck R, Lienard D, Beauduin M, Dietrich PY, Russo V, Kerger J, Masucci G, Jager E, De Greve J, Atzpodien J, Brasseur F, Coulie PG, van der Bruggen P, Boon T. Tumor regressions observed in patients with metastatic melanoma treated with an antigenic peptide encoded by gene MAGE-3 and presented by HLA-A1. Int J Cancer. 1999 Jan 18;80(2):219-30. doi: 10.1002/(sici)1097-0215(19990118)80:23.0.co;2-s. PMID 9935203
- [Background] Germeau C, Ma W, Schiavetti F, Lurquin C, Henry E, Vigneron N, Brasseur F, Lethe B, De Plaen E, Velu T, Boon T, Coulie PG. High frequency of antitumor T cells in the blood of melanoma patients before and after vaccination with tumor antigens. J Exp Med. 2005 Jan 17;201(2):241-8. doi: 10.1084/jem.20041379. PMID 15657293
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MAGE-3.A1 Peptide Mixed With CpG 7909
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The one patient who was entered into the study.
Arm/Group | MAGE-3.A1 Peptide Mixed With CpG 7909
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Detectable Cytolytic T Lymphocyte (CTL) Response Following Immunization With the MAGE-3.A1 Peptide Mixed With CpG 7909.
Description: Blood samples were collected prior to treatment and in weeks 3, 7, and 13. Specific CTL responses directed against the MAGE-3.A1 antigen were to be assessed by using restimulation in vitro, followed by staining with the A1/MAGE-3 tetramer and cloning of the tetramer-positive lymphocytes (MLPC/tetramer/cloning assay).
Time Frame: Up to 12 weeks
Population: The cytolytic T lymphocyte (CTL) response directed against the MAGE-3.A1 vaccine antigen was not analyzed due to the premature closing of this trial after only one patient was treated.
Arm/Group | MAGE-3.A1 Peptide Mixed With CpG 7909
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine the Safety of the Treatment by Measuring the Number of Patients With Dose Limiting Toxicities (DLT)
Description: All adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Scale, version 3.0.
  DLT was defined as:
  * Any Grade 3 hematological or non-hematological toxicity other than skin or flu-like symptoms.
  * Any Grade 4 toxicity. To be dose-limiting, an adverse event must be definitely, probably, or possibly related to the administration of MAGE-3.A1 peptide mixed with CpG 7909.
Time Frame: up to 12 weeks
Population: The one patient who was entered into the study and received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MAGE-3.A1 Peptide Mixed With CpG 7909
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: To Determine the Clinical Effectiveness of the Treatment by Measuring Tumor Response in Patients With Measurable Disease.
Description: Computed tomography (CT) scans were performed at screening, and at week 13. Response was assessed using RECIST version 1.0 (Therasse et al, J Natl Cancer Inst 2000; 92:205-16). Per RECIST, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions (no evaluable disease); partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria.
Time Frame: up to 12 weeks
Population: The one patient who was entered into and treated in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | MAGE-3.A1 Peptide Mixed With CpG 7909
Number analyzed (Participants) | 1
Participants
  CR | 0
  PR | 0
  SD | 0
  PD | 1

ADVERSE EVENTS:
Time Frame: up to 13 weeks
Description: All Adverse Events (AEs) occurring during the study were to be documented in the source records and on the respective AE Case Report Form (CRF), regardless of the assumption of a causal relationship. All events, which occurred after signed informed consent until end of study were documented. Toxicity was reported according to the Common Terminology Criteria for Adverse Events (CTCAE) Scale of the National Cancer Institute, version 3.0.
Arm/Group | MAGE-3.A1 Peptide Mixed With CpG 7909
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAGE-3.A1 Peptide Mixed With CpG 7909 (N=1)
Bronchitis (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 1
Influenza-like illness (General disorders) | 1
Headache (Nervous system disorders) | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Night sweats (General disorders) | 1
Injection site pain (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site scab (General disorders) | 1
Fatigue (General disorders) | 1
Weakness (General disorders) | 1

LIMITATIONS AND CAVEATS:
Study terminated due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No